CLINICAL TRIAL: NCT01736345
Title: A Study of the Communication of Genetic Test Results by Telephone: a Multi-center Study
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 29112
Record Dates: First submitted 2012-11-14; First posted 2012-11-29 (Estimated); Last update posted 2022-07-27 (Actual); Status verified 2017-07

CONDITIONS: Candidates for BRCA 1/2 Genetic Testing
MeSH Terms: interventions — Audiovisual Aids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Telephone Disclosure: Telephone Disclosure: Participants randomized to telephone disclosure will be asked to provide a personal identifier that the participant will be asked at the time of their telephone disclosure to ensure their identity.
  Interventions: Genetic: Genetic Providers; Other: Visual Aids; Other: Post-Disclosure Asessments; Other: 6 Month and 12 Month Assessments
- In Person Disclosure: Individuals opting out of randomization but still willing to participate in the research will be placed in the self-select in-person arm.
  Interventions: Genetic: Genetic Providers; Other: Visual Aids; Other: Post-Disclosure Asessments; Other: In-person Clinical Follow-Up; Other: 6 Month and 12 Month Assessments

INTERVENTIONS:
Genetic: Genetic Providers — Genetic providers (genetic counselors or nurses) will follow the standardized disclosure protocol for in-person and telephone disclosures whle completing a disclosure flow checklist.
Other: Visual Aids — Visual aids targeted to facilitate communication of genetic test results were developed based on our preliminary studies and modified based on our initial pilot study.
Other: Post-Disclosure Asessments — Within 72 hours of completion of disclosures, participants will be asked to complete post-disclosure survey again being the option to complete by the aforementioned means.
Other: In-person Clinical Follow-Up — Participants who receive their test results in person will meet with a Physician, Physician Assistant or Nurse Practitioneras part of their in person disclosure session. Participants randomiZed to telephone disclosure will be recommendedto schedule an in-person clinical follow-up appointment with a Physician, Physician Assistant or Nurse Practitioner
  Groups: In Person Disclosure
Other: 6 Month and 12 Month Assessments — At 6 months and 12 months after disclosure participants will be asked to complete survey assessments.

SUMMARY:
The overall goal of the proposed research is to evaluate psychosocial and behavioral outcomes (i.e.risks and benefits) of an innovative and efficient delivery model for genetic testing, telephone communication, as an alternative to in-person communication of genetic testing results to inform guidelines regarding the delivery of genetic information in clinical medicine.

DETAILED DESCRIPTION:
Basic science advances in genomics have provided great promise for improving human health and reducing the burden of cancer in the United States. The recent successes in genome-wide association studies (GWAS) and related technologies in identifying genetic changes associated with a variety of common diseases have fueled the rapidly growing field of personalized medicine. The promise of personalized medicine is the ability to tailor the treatment or screening of individual patients based on their genotype. Many have highlighted the urgent need for multidisciplinary translational research that focuses on how to advance gene discoveries into effective clinical applications. Genetic screening for cancer susceptibility, one application of personalized medicine, has become a standard evidence-based practice in cancer prevention. Given the complexity of genetic information and the potential social and psychological sequellae, two in-person visits (e.g. pre-test and post-test counseling) with genetic specialists are recommended for delivery of genetic testing for cancer susceptibility. With an increasing demand for genetic services, the two in-person visit delivery model presents barriers to widespread dissemination of genetic testing for disease susceptibility. Innovative delivery models for effective, efficient genetic risk communication that result in behavior change are needed. Telephone delivery of genetic services is one innovative and efficient delivery model that has the potential to expand genetic services to diverse clinical systems and address the insufficient genetic workforce as an increasing number of genetic applications enter clinical practice. While providers and patients identify advantages to telephone delivery of genetic services, they also recognize potential disadvantages particularly in the setting of a positive test result. Thus, evaluation of the psychosocial and behavioral impact of innovations to genetic service delivery (i.e. telephone communication) in diverse populations and among vulnerable subgroups are needed to optimize the health benefits, and minimize the risks of broad dissemination of clinical genetic testing for cancer susceptibility.

The goal of this research is to evaluate the psychological, behavioral and economic outcomes (i.e. risks and benefits) of an innovative and efficient delivery model of genetic services, telephone communication, as compared to the current standard, in-person communication of genetic test results. The investigators expect this research to inform evidence based practice guidelines and potentially change the paradigm of delivery of genetic services for disease susceptibility.

ELIGIBILITY:
Inclusion Criteria:

* Engligh speaking Male or Female Completed in person pretest counseling Decided to have blood drawn for clinical BRCA 1/2 Age 18 or older

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Engligh speaking Male or Female Completed in person pretest counseling Decided to have blood drawn for clinical BRCA 1/2 Age 18 or older
Sampling Method: Probability Sample
Enrollment: 289 (Actual)
Dates: Start 2012-12-03 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Number of telephone surveys completed | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Angela Bradbury, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (5):
- United States (5):
  - The John H. Stroger Jr. Hospital of Cook County, Chicago, Illinois
  - The University of Chicago, Chicago, Illinois
  - MD Anderson Cancer Center at Cooper, Camden, New Jersey
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - The Fox Chase Cancer Center, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Beri N, Patrick-Miller LJ, Egleston BL, Hall MJ, Domchek SM, Daly MB, Ganschow P, Grana G, Olopade OI, Fetzer D, Brandt A, Chambers R, Clark DF, Forman A, Gaber R, Gulden C, Horte J, Long J, Lucas T, Madaan S, Mattie K, McKenna D, Montgomery S, Nielsen S, Powers J, Rainey K, Rybak C, Savage M, Seelaus C, Stoll J, Stopfer JE, Yao XS, Bradbury AR. Preferences for in-person disclosure: Patients declining telephone disclosure characteristics and outcomes in the multicenter Communication Of GENetic Test Results by Telephone study. Clin Genet. 2019 Feb;95(2):293-301. doi: 10.1111/cge.13474. Epub 2018 Dec 7. PMID 30417332
- [Derived] Bradbury AR, Patrick-Miller LJ, Egleston BL, Hall MJ, Domchek SM, Daly MB, Ganschow P, Grana G, Olopade OI, Fetzer D, Brandt A, Chambers R, Clark DF, Forman A, Gaber R, Gulden C, Horte J, Long JM, Lucas T, Madaan S, Mattie K, McKenna D, Montgomery S, Nielsen S, Powers J, Rainey K, Rybak C, Savage M, Seelaus C, Stoll J, Stopfer JE, Yao XS. Randomized Noninferiority Trial of Telephone vs In-Person Disclosure of Germline Cancer Genetic Test Results. J Natl Cancer Inst. 2018 Sep 1;110(9):985-993. doi: 10.1093/jnci/djy015. PMID 29490071